CLINICAL TRIAL: NCT06505590
Title: STEpwise Research Program to Promote INGeniouS ONline Supportive Solutions in the Relief of Cancer-related Fatigue (STEPPING-STONe)
Brief Title: STEpwise Research Program to Promote INGeniouS ONline Supportive Solutions in the Relief of Cancer-related Fatigue
Acronym: STEPPING-STONe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: University Hospital, Bordeaux (Other); Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-A02082-43; 2023/3717 (Other: CSET number (Gustave Roussy ID))
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Cancer Diagnosis; Moderate or Severe Score of Cancer-related Fatigue (CRF)
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Educational material aid tool (Sham Comparator): Educational content on the mobile app Resilience © in the format of articles, videos or podcasts on treatment related symptoms and on validated supportive care interventions.
  Interventions: Device: Educational content
- Educational material plus self-management program - self-administered version (Experimental): Mobile app (Resilience ©) with its educational content plus a self-guided fatigue self-management program based on a cognitive behavioral therapy approach.
  Interventions: Device: Educational material plus self-management program - self-administered version
- Educational material plus self-management program - guided version with mental health professional (Experimental): Mobile app (Resilience ©) with its educational content and the self-management program of arm 2 plus weekly calls with a certified mental health professional certified in cognitive behavioural therapy for guided coaching across the self-management program.
  Interventions: Device: Educational material plus self-management program - guided version with mental health professional

INTERVENTIONS:
Device: Educational content — Patients will have access to educational content on the mobile app Resilience © in the format of articles, videos or podcasts on treatment related symptoms and on validated supportive care interventions. This version is currently public available in France and Belgium at www.resilience.care and is considered the control group (education only).
  Arms: Educational material aid tool
Device: Educational material plus self-management program - self-administered version — Patients will have access to the same mobile app (Resilience ©) with its educational content will be powered with a self-guided fatigue self-management program based on a cognitive behavioral therapy approach.
  Arms: Educational material plus self-management program - self-administered version
Device: Educational material plus self-management program - guided version with mental health professional — Patients will have access to the same mobile app (Resilience ©) with its educational content and the self-management program of arm 2 and weekly calls with a certified mental health professional certified in cognitive behavioural therapy for guided coaching across the self-management program.
  Arms: Educational material plus self-management program - guided version with mental health professional

SUMMARY:
Decentralized, randomized hybrid type 2 (effectiveness/implementation) controlled trial comparing the effectiveness of three different digital aid modalities programs in reducing the perceived burden of CRF in cancer patients while also gathering data on the implementation strategy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older.
* Having a clinical diagnosis of cancer including patients on active treatment or cancer survivors.
* Self-reporting moderate to severe CRF for at least one week (worst level of fatigue ≥ 4 on a 10-point numerical rating scale, retained in international guidelines as an optimal cutoff for identifying clinically significant CRF).
* Being able to read and understand French.
* Having access to a smartphone.
* Patients must be affiliated to a social security system or beneficiary of the same.

Exclusion Criteria:

* Suffering from current psychiatric disorder or cognitive disorder that would interfere with the ability to consent or participate.
* Currently engaging in cognitive-behavioral therapy.
* Currently engaging in another non-drug (behavioral) clinical trial.
* Suffering from physical related reversible and treatable causes of fatigue (anemia, electrolytes unbalance, infections, renal dysfunction, active metastases causing fatigue, hormonal unbalances (hypothyroidism, adrenal insufficiency, etc.) - according to physician's judgement at the moment of inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Compare the effectiveness of standard of care plus three different types of digital aid modalities for the patient. | 3 months and 6 months after the end of the program.
  Compare the effectiveness of standard of care (provided by the patient's cancer center and their treating oncologist) plus three different types of digital aid modalities for the patient (1: educational material; 2: educational material plus self-management program based on a cognitive behavioural therapy strategy - self-administered; 3: educational material plus self-management program based on a cognitive behavioural therapy strategy - guided by a psychologist) in reducing the perceived burden of CRF (cancer-related fatigue), measured as a clinically meaningful change (≥ 6 points) in fatigue scores in the fatigue subscale of the EORTC QLQ C30 questionnaire from baseline to short-term assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Franzoi MA, Pages A, Charles C, Debiasi M, Gillanders E, Ferreira A, Jacques F, Everhard S, GaryBobo G, Sambou C, Alla F, Quivy A, Morin S, Vaz-Luis I. The effectiveness and implementation of a STEpwise Program to Promote INGeniouS ONline supportive solutions for self-management of cancer-related fatigue: The STEPPING-STONe digitally enabled randomized trial. Contemp Clin Trials. 2025 Aug;155:107993. doi: 10.1016/j.cct.2025.107993. Epub 2025 Jun 26. PMID 40581251
- See also: Related Info — https://www.resilience.care/